CLINICAL TRIAL: NCT03441295
Title: Single-blind, Multi-centre, Randomized Controlled Trial Comparing Ligamys Anterior Cruciate Ligament (ACL) Repair, Internal Bracing ACL Repair and Conventional ACL Reconstruction for Relative Clinical Efficacy and Economic Benefit.
Brief Title: LIBRE (Ligamys, Internal Bracing, REconstruction) Study: Comparing Three Surgery Techniques After an Acute ACL Rupture.
Acronym: LIBRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Christiaan Heusdens, Dr., University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B300201835253; T001017N (Other Grant/Funding Number: FWO)
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Study 1 comparing Ligamys (DIS) and Internal Bracing (N=48). Study 2 comparing Internal Bracing and ACL Reconstruction (N=48).
Who Masked: Participant
Masking Description: Also the treating physiotherapist is blinded to the treatment the participant received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study 1 Ligamys (Experimental): Repair Surgery.
  Interventions: Procedure: Dynamic Intraligamentary Stabilization
- Study 1 Internal Bracing (Experimental): Repair Surgery.
  Interventions: Procedure: Internal Brace Ligament Augmentation
- Study 2 Internal Bracing (Experimental): Repair Surgery.
  Interventions: Procedure: Internal Brace Ligament Augmentation
- Study 2 Reconstruction (Active Comparator): Reconstructive Surgery.
  Interventions: Procedure: ACL Reconstruction

INTERVENTIONS:
Procedure: Dynamic Intraligamentary Stabilization — DIS, Ligamys
  Arms: Study 1 Ligamys
Procedure: Internal Brace Ligament Augmentation — IBLA
  Arms: Study 1 Internal Bracing; Study 2 Internal Bracing
Procedure: ACL Reconstruction — Conventional
  Arms: Study 2 Reconstruction

SUMMARY:
Single-blind, multi-centre, prospective, randomized controlled trial comparing Ligamys Anterior Cruciate Ligament (ACL) repair, Internal Bracing ACL repair and conventional ACL reconstruction for relative clinical efficacy and economic benefit.

Patients with a primary proximal acute ACL rupture will be included in either study 1 (0-4 weeks post rupture) or study 2 (5-12 weeks post rupture) of the LIBRE study.

DETAILED DESCRIPTION:
Rationale The conventional operative treatment of an anterior cruciate ligament (ACL) rupture is an ACL reconstruction, whereby the residual ruptured ACL is removed and replaced by an autograft hamstring tendon.

Recently, two alternative natural healing techniques have been developed and proof of concept have been established. The two repair techniques are: Dynamic Intraligamentary Stabilization (DIS) and Internal Brace Ligament Augmentation (IBLA). Both DIS and IBLA allow the rupture to heal by itself. The biggest difference between the two techniques is that the DIS system consists of a polyethylene suture and a spring screw system, which stabilizes the knee joint with the same force during flexion and extension of the knee, and the IBLA system consists of a 2mm high molecular weight polyethylene FiberTape®.

Objective The aim is to identify the optimal ACL technique for treating an acute ACL injury that can deliver an enhanced clinical efficacy and economic benefit for two time frames (0-4 weeks and 5-12 weeks) following ACL rupture.

Study design Two separate, interventional, single-blind, comparative, multi-centre, randomized controlled trials (RCTs) will be conducted. The University Hospital of Antwerp (UHA), University Hospital of Brussels (UHB) and OLV Hospital (OLVH) are the three participating sites. A total of 96 patients will be included in the study, 48 for study 1 and 48 for study 2.

The anticipated study duration is 72 months which will include a five month starting-up phase, 40 month recruitment period, a 24 month follow-up period and three months for final analysis. The study data will be collected over three periods: pre-operative, per-operative and post-operative.

To meet the aim the time-dependent nature of ACL repair surgery has to be taken into account. As the DIS should be performed within a short period after the ACL rupture, study 1 is limited to 4 weeks after ACL rupture. IBLA can be performed up to 12 weeks after ACL rupture, therefore the time limit for study 2 is 12 weeks after ACL rupture. ACL reconstruction is preferably performed when the knee has 'cooled down', and this is from 5 weeks post-rupture. There is no time limit for the ACL reconstruction, since this can be performed up to several years post-rupture.

• Study 1: RCT 1 DIS versus IBLA within 4 weeks after the ACL rupture.

• Study 2: RCT 2 IBLA versus the conventional ACL reconstruction between 5-12 weeks after the ACL rupture.

Study population Patients with a primary acute proximal ACL rupture, below the age of 50 years. The ACL remnant must be suitable for repair.

Intervention The conventional ACL reconstruction, DIS or IBLA surgery.

Main study objectives Primary outcome: Difference of 13 points in IKDC score between the reconstruction technique and the repair techniques (DIS/IBLA) 6 months postoperatively.

Main secondary outcomes: Failure/re-rupture, Tegner score, Lysholm score, EQ-5D-5L, return to work/sport, Lachman test, Pivot Shift test and complications.

Nature and extent of the burden and risks associated with participation, and benefit Proof of concept have been established and the expected complications are similar in the three treatment arms. The major benefit of the alternative repair techniques is the preservation of the native ACL and its own proprioceptors possibly leading to a faster recovery time.

ELIGIBILITY:
Inclusion Criteria:

* • Primary acute proximal ACL rupture (MRI and per-operative confirmation): 3-digit ACL rupture classification, type A (supplement 1)

  * Between 18-50 years, male or female
  * Randomization and surgery within 4 weeks after the ACL rupture (Study 1)
  * Randomization and surgery between 5-12 weeks after the ACL rupture (Study 2)
  * The ACL remnant is suitable for repair in the three treatment groups: the distal ACL remnant must be in contact with the proximal remnant/femoral condyle for at least 75% (per-operative confirmation)
  * The patient is mentally and verbally capable of participating in the study.
  * Written informed consent (according to the International Conference on Harmonisation (ICH)-GCP Guidelines).

Exclusion Criteria:

* • Known posterior cruciate ligament (PCL) and/or posterolateral ligamentous complex (PLC), lateral collateral ligament (LCL) or medial collateral ligament (MCL) grade 3 injury.

  * Known osseous fractures that could impair revalidation and/or ACL repair
  * Patients with neurological disorders or systemic diseases
  * Patients with trauma/fractures in the lower limb in the past 6 months that could influence rehabilitation
  * Non-sportive patients with a Tegner score of <3: these patients could probably counteract instability complaints with intensive physiotherapy.
  * Any inflammatory disease, Rheumatoid Arthritis (RA), Spondyloarthropathy (SpA), active malignancy
  * Patient not suited for intervention due to lack of mobility, meaning not achieving 90° of flexion before surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Score | Baseline (pre-rupture), week 13, week 26, week 52, week 104. At 6 months follow-up the primary outcome will be measured, a change of 13 IKDC points between the treatments is considered clinically meaningful.
  The International Knee Documentation Committee (IKDC) is a commonly used instrument to determine the outcome following various knee procedures, including ACL reconstructions. In essence, it is a subjective well-known tool that provides patients with an overall function score (range between 0 to 100). The score is interpreted as a measure of function with higher scores representing higher levels of function. The questionnaire addresses 3 categories: symptoms (i.e. pain, swelling, stiffness etc.), activity (rising from chair, going up and down stairs, jumping, squatting etc.) and knee function. The knee function studies focus primarily on one question: "How is the knee function post-operative compared to the situation before the injury?". In conclusion, the IKDC score is a reliable, well established and both patient and clinician friendly tool (i.e. it is easy and it requires little time to complete).

SECONDARY OUTCOMES:
Failure (re-rupture/instability complaints) | Day 1, week 2, week 6, week 13, week 26, week 52, week 104.
  Re-rupture: Clinical and MRI-confirmed. Re-rupture of the graft or the repaired ACL. Instability complaints: AP translation difference of >3 mm (Lachman test) between the injured knee and the contralateral knee and subjective instability complaints.
Tegner score | Baseline (pre-rupture), week 13, week 26, week 52, week 104.
  The Tegner (activity) score provides a method of grading daily activities, recreation, and competitive sports. It is developed to complement the Lysholm score, based on observation that a decreased activity level may hide limitations in function scores. A score is assigned based on the level of activity that the patient selects as best representing their current activity level. The final score ranges from 0 to 10, where 0 represents 'disability because of knee problems', whereas a score of 10 corresponds to 'participation in professional competitive sports'.
Lysholm score | Baseline (pre-rupture), week 13 post-operative, week 26 post-operative, week 52 post-operative, week 104 post-operative
  The Lysholm score has an easy scoring system that allows to determine an overall function score based on 8 items (pain, instability, locking, swelling, limp, stair climbing, squatting, and need for support). The total score is the sum of response to each item and ranges from 0 to 100. Higher scores indicate a better outcome with fewer symptoms or disability.
EQ-5D-5L | Baseline (pre-operative), day 1, week 2, week 6, week 13, week 26, week 52, week 104.
  EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of Health-Related Quality of Life (HRQoL). The EQ-5D consists of a descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale (score 0-100). EQ-5D-5L is an EQ-5D with 5 levels of severity for each of the 5 dimensions.
Return to work/sport | Day 1, week 2, week 6, week 13, week 26, week 52, week 104.
  Measuring after how many weeks/ post-operative the patient returns to work/sport and after how many weeks/months the patient returns to his/her pre-injury work/sport level (100% return to work/sport).
Isokinetic measurement (Biodex/CSMI) | Pre-operative, week 13, week 26, week 52.
  Isokinetic muscle torque measurements are commonly used to monitor the progress in muscle rehabilitation after knee ligament injuries. Insulated joints and their surrounding muscle groups can be tested in biomechanically correct positions, at velocities which correspond to the joint function. Various isokinetic dynamometers are in use today to evaluate muscle power such as the Biodex™ and the Computer Sports Medicine International™ (CSMI). The Biodex™ and the CSMI™ devices not only measure isometric (static) strength and concentric strength (where the muscle shortens during force production) but are also capable of measuring eccentric strength (where the muscle is lengthened while producing force). Information obtained via isokinetic measurements allows for a more efficient revalidation and evaluation of the revalidation.
MRI | Pre-operative, week 26, week 52, week 104.
  The evaluation of the healing of the ACL will be performed by means of a MRI-assessment according to Howell (Howell classification).
Visual Analogue Scale (VAS) Pain | Baseline (pre-operative), day 1, week 2, week 6, week 13, week 26, week 52, week 104.
  A VAS pain measures the amount of pain that a patient feels, ranging across a continuum from 'no pain' to 'an extreme amount of pain' (score 0-10). The distance from the 'no pain' endpoint represents the patient's pain score. VAS, is an easy assessment tool to use in patients.
Visual Analogue Scale (VAS) Satisfaction | Week 6, week 13, week 26, week 52, week 104.
  During the VAS satisfaction, patients are asked to show their satisfaction of the surgery and revalidation level on a line between 0 and 10, 0 meaning 'not satisfied' and 10 meaning 'fully satisfied' between the two endpoints of the line. The distance from the 'not satisfied' endpoint represents the patient's satisfaction score.

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Heusdens, Principal Investigator — UH, Antwerp
Locations (3):
- Belgium (3):
  - University Hospital, Antwerp, Edegem, Antwerp
  - University Hospital, Brussels, Jette, Brussels Capital
  - OLV Hospital, Aalst, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heusdens CHW, Zazulia K, Roelant E, Dossche L, van Tiggelen D, Roeykens J, Smits E, Vanlauwe J, Van Dyck P. Study protocol: a single-blind, multi-center, randomized controlled trial comparing dynamic intraligamentary stabilization, internal brace ligament augmentation and reconstruction in individuals with an acute anterior cruciate ligament rupture: LIBRƎ study. BMC Musculoskelet Disord. 2019 Nov 18;20(1):547. doi: 10.1186/s12891-019-2926-0. PMID 31739784